CLINICAL TRIAL: NCT04356248
Title: High Intensity Training and Energy Management Education vs. Standard Training and Muscle Relaxation, to Improve Quality of Life in Persons With Multiple Sclerosis, a Randomized Controlled Superiority Trial With Six Months' Follow-up
Brief Title: Training and Energy Management Education to Improve Quality of Life in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Valens (Other)
Collaborators: German Sport University, Cologne (Other); University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Jens Bansi, Principal Investigator Research and Deveopment and Sport Scientist, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-000769
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Endurance Training; Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training + energy management education (Experimental): * High-intensity interval training (HIIT): physiologically defined heart rate-controlled cycling with 80-100 rounds per minute (rpm) at 95-100% of maximum heart rate (HRmax). Participants will perform 5 × 1.5-min high-intensive exercise bouts at 95-100% of their HRmax followed by active breaks of unloaded pedalling over 2 min with the aim to achieve 60% of HRmax.
  * Energy management education (IEME): face-to-face education sessions of 6.5 h in duration over a 3-week period, all conducted by a trained occupational therapist. Participants acquire knowledge and understanding about factors that influence energy and the consequences of fatigue on their habits and lifestyle. Six weeks after returning home, the participants will receive a reinforcement letter in the form of information material to remember the content of the IEME and to reinforce the implementation of the behaviour change in managing energy.
  Interventions: Behavioral: Endurance Training; Behavioral: Education
- Low-intensity training + progressive muscle relaxation (Active Comparator): * Low-intensity training (ST): participants will exercise for 24 min continuously at 65% of participants' HRmax (60-70 rpm).
  * Progressive muscle relaxation (PMR): The aim of PMR is to achieve enhanced mental relaxation by reducing muscle tension. Participants will attend six 1-h group sessions over the 3-week intervention period, instructed by a trained physical therapist. Six weeks after returning home, the participants will receive a reinforcement letter with information material for remembering the content of the PMR techniques and to reinforce the implementation of the exercises at home.
  Interventions: Behavioral: Endurance Training; Behavioral: Education

INTERVENTIONS:
Behavioral: Endurance Training — Treatment in both arms consists of specific endurance exercise modalities (HIIT or ST). Treatments differ in the applied training intensities. Participants in both arms will exercise 3 times per week over a period of 3 weeks on a bicycle ergometer. Exercise sessions will be supervised by a trained physical therapist. Exercise intensity will be heart rate monitored based on the maximum heart rate (HRmax) assessed during the initial cardiopulmonary exercise test. Exercise sessions in both arms will include a warm-up and a cool-down period at low intensity (50% HRmax) for 3 min each.
Behavioral: Education — Treatment in both arms consists of specific energy management education interventions (IEME or PMR). Treatments differ in the applied education approaches. Participants in both arms will exercise 2 times per week over a period of 3 weeks.

SUMMARY:
Persons with Multiple Sclerosis (PwMS) often suffer from impaired mobility and reduced aerobic capacity. Moreover, 65% of PwMS recognize fatigue as their most disabling symptom that quickly impacts patients' health-related quality of life (QoL). Systematic reviews that evaluate therapeutic options for MS-neurorehabilitation show good evidence for exercise and energy management/conservation programs to improve fatigue or its impact on daily life. Guidelines recommend a multidisciplinary approach but to date only unimodal interventions are investigated. This study aims to investigate the influence of the combination of two different therapeutic concepts: inpatient energy management education (IEME) + High-intensity interval training (HIIT). This intervention is compared with a control group that undergoes progressive muscle relaxation (PMR) + low-intensity training (ST). IEME or PMR is performed on two days (tue-thur) and HIIT or ST on three days (mo-wed-fr) / week. The primary outcome is the effect on the quality of life after three weeks rehabilitation and after returning home (at 4 and 6 months follow-up) in PwMS.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis (revised McDonald criteria, 2018).
* Age >18y
* Expanded Disability Status Scale (EDSS) score ≤ 6.5
* Fatigue Scale of Motor and Cognitive function (FSMC) total score > 43
* Literacy and understanding German
* Informed Consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding / have the intention to become pregnant during the course of the study
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Cognitive impairment Mini-Mental State Examination (MMSE) < 21
* Major Depression or Hospital Anxiety and Depression Scale (HADS) >11 at baseline
* Stem cell treatment in the last 6 months
* Participation in a previous high-intensity interval training (HIIT) or inpatient energy management education (IEME) study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Short-form 36 (SF-36) | 6 months (day 0 - day 183) with time points set after three weeks (day 21) and 4 months (day 122).
  Changes of health-related quality of life will be assessed with the SF-36. The SF-36 questionnaire comprises 36 items. Scores range from 0 to 100 with higher values indicating better QoL.

SECONDARY OUTCOMES:
Indicators of inflammatory activity | Three weeks (day 0 - day 21).
  Soluble factors that are known to be produced or secreted in response to exercise and are suspected to modify immune homeostasis and blood brain barrier function through their inflammatory and anti-inflammatory properties. Changes of Matrix-metalloproteinases-2 (MMP-2), Tryptophan, Kynurenine, Kynurenine acid, Interferon-gamma (IFN-Gamma) and Interleukin-6 (IL-6) will be assessed. Higher values indicate higher levels of Inflammation.
Cardiorespiratory Fitness | Three weeks (day 0 - day 21).
  Changes of cardiorespiratory fitness will be measured by peak oxygen consumption achieved in the cardiopulmonary exercise test. Higher values indicate better cardiorespiratory fitness.
Self-efficacy in performing energy conservation strategies (SEPECSA) | Six months (day 0 - day 183) with time points set after three weeks (day 21) and after 4 months (day 122).
  Changes of self-efficacy in performing energy conservation strategies will be assessed with a self-reported questionnaire. The questionnaire consists of 14 items. The participants are asked to rank how confident they are that they can perform each item on a scale from 1 (= not at all confident/sure) to 10 (= completely confident/sure). The final score is found by adding the total items' score and dividing it by 14, with higher scores indicating greater confidence in self-efficacy.
Self-perceived competence in activities of daily living (OSA) | Six months (day 0 - day 21) with time points set after three weeks (day 21) and four months (day 122).
  Changes of self-perceived competence are assessed with a self reported questionnaire. The questionnaire consists of 21 items that represent participation in habits and roles, performance of skills, and volition for participation. Participants rate each item with two 4-point likert scales to indicate their self-perception of occupational competence (I have a lot of problems doing this - I have some difficulty doing this - I do this well - I do this extremely well) and value for importance (This is not so important to me - This is important to me - This is more important to me - This is most important to me). Following these two steps, clients review their ratings and choose areas of occupational performance and participation that they would like to change. Higher scores indicate better competences.
Fatigue Scale of motor and cognitive function (FSMC) | Six months (day 0 - day 183) with time points set after three weeks (day 21) and four months (day 122).
  Changes of motor and cognitive fatigue are assessed on a 5-point likert-scale. Max 50 Points for subscales, 100 Points for the Total score. Cut-off for fatigue is set for the total score at 43 and for the motoric and cognitive subscores at 22 with higher values participants being more fatigued.
Hospital Anxiety and Depression Scale (HADS) | 6 months (day 0 - day 183) with time points set after three weeks (day 21) and four months (day 122).
  Changes of anxiety and depression over three weeks training on a 4-point likert scale scored 0-3. Max 21 Points for each subscale, cut off for anxiety and Depression are set at 7 Points higher values represent more anxiety and Depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bansi, PhD, Principal Investigator — Klinik Valens
Locations (1):
- Kliniken-Valens, Valens, Canton of St. Gallen, Switzerland

REFERENCES:
- [Derived] Kupjetz M, Langeskov-Christensen M, Riemenschneider M, Inerle S, Ligges U, Gaemelke T, Patt N, Bansi J, Gonzenbach RR, Reuter M, Rosenberger F, Meyer T, McCann A, Ueland PM, Eskildsen SF, Nygaard MKE, Joisten N, Hvid L, Dalgas U, Zimmer P. Persons With Multiple Sclerosis Reveal Distinct Kynurenine Pathway Metabolite Patterns: A Multinational Cross-Sectional Study. Neurol Neuroimmunol Neuroinflamm. 2025 Nov;12(6):e200461. doi: 10.1212/NXI.0000000000200461. Epub 2025 Sep 18. PMID 40966534
- [Derived] Belen S, Patt N, Kupjetz M, Ueland PM, McCann A, Gonzenbach R, Bansi J, Zimmer P. Vitamin B6 status is related to disease severity and modulated by endurance exercise in individuals with multiple sclerosis: a secondary analysis of a randomized controlled trial. Am J Clin Nutr. 2025 Jun;121(6):1403-1414. doi: 10.1016/j.ajcnut.2025.04.014. Epub 2025 Apr 17. PMID 40252731
- [Derived] Kupjetz M, Patt N, Joisten N, Ueland PM, McCann A, Gonzenbach R, Bansi J, Zimmer P. Baseline Inflammation but not Exercise Modality Impacts Exercise-induced Kynurenine Pathway Modulation in Persons With Multiple Sclerosis: Secondary Results From a Randomized Controlled Trial. Int J Tryptophan Res. 2024 Nov 11;17:11786469241284423. doi: 10.1177/11786469241284423. eCollection 2024. PMID 39534856
- [Derived] Kupjetz M, Patt N, Joisten N, Ueland PM, McCann A, Gonzenbach R, Bansi J, Zimmer P. The serum kynurenine pathway metabolic profile is associated with overweight and obesity in multiple sclerosis. Mult Scler Relat Disord. 2023 Apr;72:104592. doi: 10.1016/j.msard.2023.104592. Epub 2023 Mar 1. PMID 36881945
- [Derived] Patt N, Kool J, Hersche R, Oberste M, Walzik D, Joisten N, Caminada D, Ferrara F, Gonzenbach R, Nigg CR, Kamm CP, Zimmer P, Bansi J. High-intensity interval training and energy management education, compared with moderate continuous training and progressive muscle relaxation, for improving health-related quality of life in persons with multiple sclerosis: study protocol of a randomized controlled superiority trial with six months' follow-up. BMC Neurol. 2021 Feb 11;21(1):65. doi: 10.1186/s12883-021-02084-0. PMID 33573608